CLINICAL TRIAL: NCT05340894
Title: A Randomaized ,Double Study ,Aims to Compare Between Mckenzie and William's Exercises in Order to Find Which Method Has Better Effect on Adolescents With Non Specific Low Back Pain
Brief Title: Mckenzie Versus William Exercise for Non Specific Low Back Pain in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham Hany Mohamed Mahmoued Elmahdy, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003327
Record Dates: First submitted 2022-03-15; First posted 2022-04-22 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-08

CONDITIONS: Non Specific Low Back Pain
Keywords: Adolescents, Balance, Low Back Pain, McKenzie Exercises, and William's Exercises.
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mckenzie group (Active Comparator): * adolescents will receive 4 weeks Mckenzie exercise program
  * Follow-up:pre-test (Baseline), 2 weeks post-test and 4 weeks post-test.
  Interventions: Procedure: MCKENZIE exercises
- William's group (Active Comparator): * adolescents will receive 4 weeks William's exercise program
  * Follow-up:pre-test (Baseline), 2 weeks post-test and 4 weeks post-test.
  Interventions: Procedure: WILLIAM'S exercises

INTERVENTIONS:
Procedure: MCKENZIE exercises — McKenzie method is popular amongst physiotherapists as a management approach for spinal pain and McKenzie exercises for LBP are beneficial treatment for increasing flexibility of spine and improving the pain with better results in pain relief
  Arms: Mckenzie group
Procedure: WILLIAM'S exercises — William flexion exercise is to reduce pain or soreness and provide lower trunk stability by actively developing the abdominal muscles,gluteus maximus and hamstring, passively stretching the hip flexors and lower back muscles(sacro spinalis) and to restore or improve the work balance between the postural flexor and extensor muscle groups
  Arms: William's group

SUMMARY:
MCKENZIE EXERCISE VERSUS WILLIAMS EXERCISE ON DECREASING PAIN IN ADOLESCENT WITH NON SPECIFIC LOW BACK PAIN

Low back pain is uncommon in the first decade of life,but prevalence increases steeply during the teenage years; around 40% of 9-18-year olds in high-income, medium-income, and low-income countries report having had low back pain. NSLBP represents about 85% of LBP patients seen in primary care. Non-specific low back pain is one of the most common health problems and is the leading cause of disability in young adults. During school age, the overall risk of low back pain is similar to adults, with prevalence rates as high as 70% to 80% by the age of 20 years old Non-specific low back pain is defined as low back pain not attributable to a recognisable, known specific pathology.

Understanding back pain in adolescents is crucial to obtain timely diagnosis and determine appropriate treatment. Proper treatment and management of LBP in the adolescent years can minimize back pain lasting into adulthood Non pharmacological treatments are emphasised over pharmacological interventions in the management of persistent non-specific low back pain.

natinal institute for health and care excellence(NICE) 2016 draft guideline endorses self-management, exercise, manual therapy, psychological therapies, combined physical and psychological programmes, return-to-work programmes, and radiofrequency denervation.

Back exercises can be an inexpensive and easy option of treatment for NSLBP and proven to be effective. McKenzie extension exercise and William flexion exercise are the most common types of back exercises.

Selection the appropriate treatment method is important. So this study will be aimed to compare between Mckenzie and William's exercises in order to find which method has better effect on adolescents with NSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 14 to 18 years.
* Diagnosed as non-specific low back pain.
* Medically and clinically stable.
* All participants are within normal range weight and height.

Exclusion Criteria:

Adolescents have one or more of the followings will be excluded:

* Any spinal deformities.
* History of spinal or pelvic surgery.
* Specific spinal pathologies as cauda equina syndrome, cord compression, infection, fracture, neoplasm, inflammatory disease, whiplash associated disorders and vertebro-basilar insufficiency.
* Any visual or auditory problems that interfere with the rehabilitation program.
* Children with significant mental or psychological problems that interfere with understanding instructions.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — adolescents male only
Enrollment: 30 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | changes in pain at 4 weeks
  This will be used to determine the intensity of pain.The VAS is a valid and reliable measure of chronic pain intensity . It is the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. Operationally, a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end The patient will mark on the line at the point that he feels which represents his perception of the current state.The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the child marks .

SECONDARY OUTCOMES:
ModifiedSchober's Test(MSchober test) | changes in back flexibility in 4 weeks
  The mSchober test is frequently used method for assessing lumbar flexion range of motion (ROM).
  Test will be done as follows:
  * The participant will stand in neutral erect position without shoes.
  * The assessor will marks 1 point 5 cm below and 1 point 10 cm above the lumbosacral junction(dimples of Venus), that is, 15 cm in upright position.
  * The participant will be asked to make 2 attempts to bend forward as far as possible, the first will be a trial attempt, and the assessor measured the distance between the marks on the second attempt
  * The increase in distance between the marks was then calculated as the measure of lumbar flexion ROM.
  * In general, the measure should increase by at least 6 cm to 21 cm. An increase of less than 6 cm suggests decreased lumbar spinal mobility.

OTHER OUTCOMES:
YMED TEST Balance Test | changes in balance in 4 weeks
  This smart phone application was developed by Physio tools YMED; a group from the kwangju Health College, South Korea. It allows the performance of several tests: vestibular balance test, sitting balance test, knee balance test and board balance test .
  Vestibular and board balance tests will be used as the following:
  • Vestibular balance test: Smart phone device will be fixed on the patient's back by strap and he will be asked firstly to keep standing with open eyes for 10 seconds and therapist click start button then to keep standing with closed eyes for 10 seconds and wait for report of test.
  • Board balance test: Patient will be asked to stand on a balance board and fix the smart phone on the board and the patient will be asked to stand steady as much as can for 10 seconds then print the reports.